CLINICAL TRIAL: NCT04426851
Title: Investigation of Pharmacokinetics and Absolute Bioavailability of BI 1358894 Administered Orally as Tablet Co-administered With an Intravenous Microtracer Dose of [C-14]-BI 1358894 in Healthy Male Volunteers Via a Non-randomised, Open-label, Fixed-sequence Trial (Part 1) Followed by a Randomised, Open-label, Single-dose, Two-period, Two-sequence Cross-over Relative Bioavailability Trial in BI 1358894 Oral Suspension (Part 2)
Brief Title: A Study in Healthy Men to Test How BI 1358894 is Taken up in the Body and How Food Influences the Amount of BI 1358894 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1402-0016; 2020-000351-13 (EudraCT Number)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — TRPC inhibitor BI 1358894; Carbon-14

STUDY DESIGN:
Intervention Model Description: Part 1: non-randomized, fixed-sequence design Part 2: randomized, two-period, two-sequence, crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1358894: Part 1: tablet (T1) - (C14) i.v (R1), Part 2: fasted (R2) - fed (T2) (Experimental): BI 1358894
  Interventions: Drug: BI 1358894; Drug: BI 1358894 (C-14) intravenous solution
- BI 1358894: Part 1: tablet (T1) - (C14) i.v (R1), Part 2: fed (T2) - fasted (R2) (Experimental): BI 1358894
  Interventions: Drug: BI 1358894; Drug: BI 1358894 (C-14) intravenous solution

INTERVENTIONS:
Drug: BI 1358894 — Tablet
Drug: BI 1358894 (C-14) intravenous solution — BI 1358894 mixed with [carbon labelled (C-14)] BI 1358894
Drug: BI 1358894 — Oral suspension

SUMMARY:
The main objective of Part 1 of this trial is to investigate the absolute bioavailability of BI 1358894 with an intravenous microdose formulation containing labelled [C-14] BI 1358894 and an unlabelled oral tablet formulation of BI 1358894 in healthy male subjects.

The main objective of Part 2 of this trial is to investigate the relative bioavailability of BI 1358894 administered as an oral suspension.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
* Male subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 90 days after trial completion:
* Use of adequate contraception of the female partner, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device that started at least 2 months prior to first study drug administration or barrier method (e.g. diaphragm with spermicide) or,
* Sexually abstinent or
* A vasectomy performed at least 1 year prior to screening (with medical assessment of the surgical success) or
* Surgically sterilised female partner (including hysterectomy, bilateral tubal occlusion or bilateral oophorectomy) or
* Postmenopausal female partner, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with FSH (follicle stimulating hormone) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 40 to 100 bpm
* C-reactive protein (CRP) > upper limit of normal (ULN), liver or kidney parameter above ULN
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase I trial which investigated the pharmacokinetics and absolute bioavailability of BI 1358894 administered orally as tablet co-administered with an intravenous microtracer dose of labelled [C-14]-BI 1358894 in healthy male volunteers via a non-randomised, open-label, fixed-sequence trial (part 1) followed by a randomised, openlabel, single-dose, two-period, two-sequence cross-over relative bioavailability trial in BI 1358894 oral suspension (part 2).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 1358894: Part 1: Tablet (T1) - (C14) i.v (R1), Part 2: Fasted (R2) - Fed (T2): In Part 1: Period 1 of the study participants received on Day 1 one single oral dose of two 50 milligram (mg) BI 1358894 tablets (total dose=100mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) (Test 1-T1). 5 hours after the oral administration (i.e. at the time of the expected tmax) participants received one single dose of 10 mL intravenous (i.v) infusion of 100 microgram (µg) BI 1358894 using a mixture of 90 µg unlabelled and 10 µg [C-14] labelled BI 1358894 (Reference 1-R1).
  After 15 days of washout the Part 2: Period 2 of the study started and participants received on Day 1 of Period 2 one single dose of 100 mg BI 1358894 administered as an oral suspension with 240 mL of water after an overnight fast of at least 10 h when fasted (Reference 2-R2). After 17 days of washout Part 2: Period 3 started and participants received on Day 1 of Period 3 one single dose 100 mg BI 1358894 administered as an oral suspension with 240 mL of water following a high-fat, high-calorie breakfast when fed (Test 2-T2).
- BI 1358894: Part 1: Tablet (T1) - (C14) i.v (R1), Part 2: Fed (T2) - Fasted (R2): In Part 1: Period 1 of the study participants received on Day 1 one single oral dose of two 50 milligram (mg) BI 1358894 tablets (total dose=100mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) (Test 1-T1). 5 hours after the oral administration (i.e. at the time of the expected tmax) participants received one single dose of 10 mL intravenous (i.v) infusion of 100 microgram (µg) BI 1358894 using a mixture of 90 µg unlabelled and 10 µg [C-14] labelled BI 1358894 (Reference 1-R1).
  After 15 days of washout Part 2: Period 2 started and participants received on Day 1 of Period 2 one single dose 100 mg BI 1358894 administered as an oral suspension with 240 mL of water following a high-fat, high-calorie breakfast when fed (Test 2-T2). After 17 days of washout the Part 2: Period 3 of the study started and participants received on Day 1 of Period 3 one single dose of 100 mg BI 1358894 administered as an oral suspension with 240 mL of water after an overnight fast of at least 10 h when fasted (Reference 2-R2).
Period: Part 1: Period 1+Washout
Arm/Group | BI 1358894: Part 1: Tablet (T1) - (C14) i.v (R1), Part 2: Fasted (R2) - Fed (T2) | BI 1358894: Part 1: Tablet (T1) - (C14) i.v (R1), Part 2: Fed (T2) - Fasted (R2)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Part 2: Period 2+Washout
Arm/Group | BI 1358894: Part 1: Tablet (T1) - (C14) i.v (R1), Part 2: Fasted (R2) - Fed (T2) | BI 1358894: Part 1: Tablet (T1) - (C14) i.v (R1), Part 2: Fed (T2) - Fasted (R2)
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 0
Period: Part 2: Period 3+Washout
Arm/Group | BI 1358894: Part 1: Tablet (T1) - (C14) i.v (R1), Part 2: Fasted (R2) - Fed (T2) | BI 1358894: Part 1: Tablet (T1) - (C14) i.v (R1), Part 2: Fed (T2) - Fasted (R2)
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all subjects who were randomized and treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1358894: Part 1: Tablet (T1) - (C14) i.v (R1), Part 2: Fasted (R2) - Fed (T2) | BI 1358894: Part 1: Tablet (T1) - (C14) i.v (R1), Part 2: Fed (T2) - Fasted (R2) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.2 (11.9) | 37.8 (14.0) | 38.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Concentration-time Curve of BI 1358894 Over the Time Interval From 0 to Infinity After i.v. Administration and After Oral Administration (AUC0-infinity)
Description: Area under the concentration-time curve of BI 1358894 over the time interval from 0 to infinity after i.v. administration and after oral administration (AUC0-infinity) is reported. The values were calculated using the Analysis of variance (ANOVA) model which included effects accounting for the following sources of variation: 'subjects' and 'formulation'. The effect 'subjects' was considered as random, whereas 'formulation' was considered as fixed.
  Standard error is actually geometric standard error. Time Frame: For "BI 1358894 (C-14) 100 ug i.v" samples were collected at 5h, 5.083, 5.16, 5.25, 5.5, 5.75, 6, 6.5, 7,8, 10, 12, 24, 34, 48, 72, 96, 144, 192, 240, 312 h after oral dose of BI 1358894 on Day 1 of Period 1.
Time Frame: Within 2 hours (h) before and at 15 minutes (min), 30 min, 1 h, 1.5, 2, 3, 4, 5, 5.083, 5.16, 5.25, 5.5, 5.75, 6, 6.5, 7,8, 10, 12, 24, 34, 48, 72, 96, 144, 192, 240, 312 h after oral dose of BI 1358894 on Day 1 of Period 1. Continues in description.
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects in the TS who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS even if he contributed only 1 PK parameter value for 1 period to the statistical assessment. Descriptive and model-based analyses of PK parameters were based on the PKS.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*millimol/Liter/kilogram
Groups:
- BI 1358894 100 mg Tablet Fasted: On Day 1 of Part1: Period 1 participants received one single oral dose of two 50 milligram (mg) BI 1358894 tablets (total dose=100mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) (Test 1-T1).
- BI 1358894 (C-14) 100 ug i.v: Participants received on Day 1 of Part 1: Period 1 one single dose of 10 mL intravenous (i.v) infusion of 100 microgram (µg) BI 1358894 using a mixture of 90 µg unlabelled and 10 µg [C-14] labelled BI 1358894 (Reference 1-R1). The i.v infusion started 5 hours after the administration of Test 1-T1.
Arm/Group | BI 1358894 100 mg Tablet Fasted | BI 1358894 (C-14) 100 ug i.v
Number analyzed (Participants) | 12 | 12
hour*millimol/Liter/kilogram | 96 (NA) — Adjusted geometric standard error=1.093 | 209 (NA) — Adjusted geometric standard error=1.093
Statistical Analysis 1: Comparison: BI 1358894 100 mg Tablet Fasted vs BI 1358894 (C-14) 100 ug i.v; The Analysis of variance (ANOVA) model included effects accounting for the following sources of variation: 'subjects' and 'formulation'. The effect 'subjects' was considered as random, whereas 'formulation' was considered as fixed; Test type: Other; Ratio of the geometric means (%) = 45.9, 90% CI 2-sided [41.4 to 50.9] — Ratio was calculated as: BI 1358894 100 mg tablet fasted/BI 1358894 (C-14) 100 ug i.v. Intra-individual geometric coefficient of variation (gCV)=14.3

2. Primary Outcome: Part 2: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 to 312 h (AUC 0-312)
Description: Area under the concentration-time curve of BI 1358894 in plasma over the time interval from 0 to 312 h (AUC 0-312) is reported. The values were calculated using the Analysis of variance (ANOVA) model which included effects accounting for the following sources of variation: 'sequence or block', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. Standard error is actually geometric standard error.
Time Frame: Within 2 hours (h) before drug administration and at 15 minutes (min), 30 min, 1 h, 1.5, 2, 3, 4, 5, 6, 7,8, 10, 12, 24, 34, 48, 72, 96, 144, 192, 240, 312 h after administration of BI 1358894.
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects in the TS who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS even if he contributed only 1 PK parameter value for 1 period to the statistical assessment. For both arms 11 subjects were treated.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour* nanomol/Liter (h*nmol/L)
Groups:
- BI 1358894 100 mg Oral Suspension Fasted: Participants received one single dose of 100 milligram (mg) BI 1358894 administered as an oral suspension with 240 milliliter (mL) of water after an overnight fast of at least 10 hours when fasted (Reference 2-R2).
- BI 1358894 100 mg Oral Suspension Fed: Participants received one single dose of 100 milligram (mg) of BI 1358894 administered as an oral suspension with 240 milliliter (mL) of water following a high-fat, high-calorie breakfast when fed (Test 2-T2).
Arm/Group | BI 1358894 100 mg Oral Suspension Fasted | BI 1358894 100 mg Oral Suspension Fed
Number analyzed (Participants) | 11 | 11
hour* nanomol/Liter (h*nmol/L) | 12217 (NA) — Adjusted geometric standard error = 1.080 | 17271 (NA) — Adjusted geometric standard error = 1.080
Statistical Analysis 1: Comparison: BI 1358894 100 mg Oral Suspension Fasted vs BI 1358894 100 mg Oral Suspension Fed; The ANOVA model included effects accounting for the following sources of variation: 'sequence or block', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; Ratio of the geometric means (%) = 141.4, 90% CI 2-sided [129.3 to 154.6] — Ratio was calculated as: BI 1358894 100 mg oral suspension fed/BI 1358894 100 mg oral suspension fasted. Intra -individual geometric coefficient of variation (gCV)=10.9

3. Secondary Outcome: Part 1: Maximum Measured Concentration of BI 1358894 in Plasma After i.v. Administration and After Oral Administration (Cmax)
Description: Maximum measured concentration of BI 1358894 in plasma after i.v. administration and after oral administration(Cmax) is reported.
  Time Frame: For "BI 1358894 (C-14) 100 ug i.v" samples were collected at 5h, 5.083, 5.16, 5.25, 5.5, 5.75, 6, 6.5, 7,8, 10, 12, 24, 34, 48, 72, 96, 144, 192, 240, 312 h after oral dose of BI 1358894 on Day 1 of Period 1.
Time Frame: Within 2 hours before and at 15 minutes (min), 30 min, 1 hour (h), 1.5, 2, 3, 4, 5, 5.083, 5.16, 5.25, 5.5, 5.75, 6, 6.5, 7,8, 10, 12, 24, 34, 48, 72, 96, 144, 192, 240, 312 h after oral dose of BI 1358894 on Day 1 of Period 1. Continues in description.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/Liter (nmol/L)
Arm/Group | BI 1358894 100 mg Tablet Fasted | BI 1358894 (C-14) 100 ug i.v
Number analyzed (Participants) | 12 | 12
nanomol/Liter (nmol/L) | 408 (34.1) | 0.847 (28.8)

4. Secondary Outcome: Part 2: Maximum Measured Concentration of BI 1358894 in Plasma After Administration of the Oral Suspension (Cmax)
Description: Maximum measured concentration of BI 1358894 in plasma after administration of the oral suspension (Cmax) is reported. The Analysis of variance (ANOVA) model included effects accounting for the following sources of variation: 'sequence or block', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. Standard error is actually geometric standard error.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomol/Liter (nmol/L)
Arm/Group | BI 1358894 100 mg Oral Suspension Fasted | BI 1358894 100 mg Oral Suspension Fed
Number analyzed (Participants) | 11 | 11
nanomol/Liter (nmol/L) | 810 (NA) — Adjusted geometric standard error = 1.082 | 529 (NA) — Adjusted geometric standard error = 1.082
Statistical Analysis 1: Comparison: BI 1358894 100 mg Oral Suspension Fasted vs BI 1358894 100 mg Oral Suspension Fed; [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio of the geometric means (%) = 65.3, 90% CI 2-sided [54.6 to 78.0] — Ratio was calculated as: BI 1358894 100 mg oral suspension fed/BI 1358894 100 mg oral suspension fasted. Intra - individual geometric coefficient of variation (gCV)=22.5

5. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 Extrapolated to Infinity After Administration of the Oral Suspension (AUC0-infinity)
Description: Area under the concentration-time curve of BI 1358894 in plasma over the time interval from 0 extrapolated to infinity after administration of the oral suspension (AUC0-infinity) is reported. The Analysis of variance (ANOVA) model included effects accounting for the following sources of variation: 'sequence or block', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. Standard error is actually geometric standard error.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomol/Liter (h*nmol/L)
Arm/Group | BI 1358894 100 mg Oral Suspension Fasted | BI 1358894 100 mg Oral Suspension Fed
Number analyzed (Participants) | 11 | 11
hour*nanomol/Liter (h*nmol/L) | 13510 (NA) — Adjusted geometric standard error = 1.086 | 20052 (NA) — Adjusted geometric standard error = 1.086
Statistical Analysis 1: Comparison: BI 1358894 100 mg Oral Suspension Fasted vs BI 1358894 100 mg Oral Suspension Fed; [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio of the geometric means (%) = 148.4, 90% CI 2-sided [138.1 to 159.5] — Ratio was calculated as: BI 1358894 100 mg oral suspension fed/BI 1358894 100 mg oral suspension fasted. Intra - individual geometric coefficient of variation (gCV) =8.7

ADVERSE EVENTS:
Time Frame: BI tablet = From treatment start until start of C14, up to 1 day. BI fed, BI fasted and BI C14 = day of treatment + 11 days Residual Effect Period (REP), up to 12 days.
Description: Treated set (TS): The treated set includes all subjects who were randomized and treated with at least one dose of study drug.
Groups:
- BI 1358894 100 mg Tablet Fasted: Participants received on Day 1 of Part 1: Period 1 one single oral dose of two 50 milligram (mg) BI 1358894 tablets (total dose=100mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) (Test 1-T1).
Arm/Group | BI 1358894 100 mg Tablet Fasted | BI 1358894 (C-14) 100 ug i.v | BI 1358894 100 mg Oral Suspension Fasted | BI 1358894 100 mg Oral Suspension Fed
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 6/12 | 9/12 | 6/11 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1358894 100 mg Tablet Fasted (N=12) | BI 1358894 (C-14) 100 ug i.v (N=12) | BI 1358894 100 mg Oral Suspension Fasted (N=11) | BI 1358894 100 mg Oral Suspension Fed (N=11)
Headache (Nervous system disorders) | 5 | 5 | 5 | 7
Somnolence (Nervous system disorders) | 0 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 0
Catheter site haematoma (General disorders) | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT04426851/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT04426851/SAP_001.pdf